CLINICAL TRIAL: NCT04761003
Title: Efficacy And Safety Of Thoracoscopic Cryobiopsy In Patients With Undiagnosed Exudative Pleural Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tamer Awad, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Thoracoscopic cryobiopsy
Record Dates: First submitted 2021-02-14; First posted 2021-02-18 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Pleura; Exudate

STUDY DESIGN:
Intervention Model Description: A full medical history was obtained. Medical history, clinical examination and local chest examination for signs of pleural effusion, Radiological data include chest X-ray, chest computed tomography (CT), and chest ultrasound (US) for localization of a better entry site.
  Thoracoscopy procedure the procedure was performed in the lateral decubitus position with the affected side upward under conscious sedation. Local anesthesia consisting of 2% lignocaine was administered to the skin, subcutaneous tissue, muscle, and parietal pleura.
  The appearance of the parietal and visceral pleural was assessed and recorded. Pleural biopsies were obtained using rigid forceps and cryoprobe during rigid medical thoracoscopy Complications during thoracoscopy were recorded as bleeding and surgical emphysema.
  Samples were directly fixed in 10% formalin solution Biopsies obtained were examined pathologically with stress on size and quality of the sample.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Cryobiopsy group): (Active Comparator): patients where patients will be subjected to thoracoscopic cryobiopsy.
  Interventions: Device: Thoracoscopy forceps
- Group II (Forceps group) (Active Comparator): patients where patients will be subjected to thoracoscopic forceps biopsy.
  Interventions: Device: Thoracoscopy forceps

INTERVENTIONS:
Device: Thoracoscopy forceps — take pleural biopsy
  Other Names: Thoracoscopic cryobiopsy

SUMMARY:
To demonstrated the efficacy and safety of taking biopsy specimens from parietal pleura in undiagnosed exudative pleural effusion

DETAILED DESCRIPTION:
Pleural effusions are either transudate or exudate according to the biochemical analysis of aspirated pleural fluid. Thoracentesis or blind pleural biopsy may not provide a definitive diagnosis. Cryobiopsy has more successful diagnostic results than forceps biopsies with complications (only hemorrhage) during procedures. Cryobiopsy can obtain more diagnostic biopsies due to the size of the biopsies and best property in expressions of an artifact-free sample area

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as exudative pleural effusion according to Light criteria .informed written consents were taken from all patients enrolled in the study

Exclusion Criteria:

* patients who refused participation ,patients unfit for medical thoracoscopy (MT) will be excluded from the study such as:Uncooperative patient ,Severe uncorrected hypoxemia in spite of continuous oxygen administration, because it's necessary to keep oxygen saturation above 90 % during procedure ,patients who could not tolerate the lateral decubitus position for a period long adequate to do the thoracoscopy, unstable cardiovascular or hemodynamic condition, uncorrected Coagulation defects and small pleural space

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
efficacy which determined by the diagnostic yield | baseline
  comparing forceps biopsy and cryobiopsy as regard: efficacy which determined by the diagnostic yield.
efficacy which determined by the size of biopsy | baseline
  comparing forceps biopsy and cryobiopsy as regard: efficacy which determined by the size of biopsy.
The incidence of complications | baseline
  comparing forceps biopsy and cryobiopsy as regard: Safety which determined by the incidence of complications

CONTACTS AND LOCATIONS:
Overall Officials: Raed E ALI, MD, Study Chair — Mansoura University; Ahmed E Mansour, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Result] Light RW. Pleural diseases. Curr Opin Pulm Med. 2003 Jul;9(4):251-3. doi: 10.1097/00063198-200307000-00001. No abstract available. PMID 12806235
- [Result] Noppen M. The utility of thoracoscopy in the diagnosis and management of pleural disease. Semin Respir Crit Care Med. 2010 Dec;31(6):751-9. doi: 10.1055/s-0030-1269835. Epub 2011 Jan 6. PMID 21213207
- [Result] Porcel JM. Pleural fluid biomarkers: beyond the Light criteria. Clin Chest Med. 2013 Mar;34(1):27-37. doi: 10.1016/j.ccm.2012.11.002. Epub 2013 Jan 17. PMID 23411054
- [Result] Tousheed SZ, Manjunath PH, Chandrasekar S, Murali Mohan BV, Kumar H, Hibare KR, Ramanjaneya R. Cryobiopsy of the Pleura: An Improved Diagnostic Tool. J Bronchology Interv Pulmonol. 2018 Jan;25(1):37-41. doi: 10.1097/LBR.0000000000000444. PMID 29261578
- [Result] Bonniot JP, Homasson JP, Roden SL, Angebault ML, Renault PC. Pleural and lung cryobiopsies during thoracoscopy. Chest. 1989 Mar;95(3):492-3. doi: 10.1378/chest.95.3.492. PMID 2920573
- [Result] Hetzel J, Hetzel M, Hasel C, Moeller P, Babiak A. Old meets modern: the use of traditional cryoprobes in the age of molecular biology. Respiration. 2008;76(2):193-7. doi: 10.1159/000135934. Epub 2008 Jun 26. PMID 18708736
- [Result] Porcel JM, Light RW. Diagnostic approach to pleural effusion in adults. Am Fam Physician. 2006 Apr 1;73(7):1211-20. PMID 16623208